CLINICAL TRIAL: NCT03188952
Title: Validity of International Caries Classification and Management System (ICCMS) Versus International Caries Detection and Assessment System (ICDAS ) in Caries Assessment : Invivo Diagnostic Study
Brief Title: Validity of ICDAS Versus ICCMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, amr sobhy, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: oper206
Record Dates: First submitted 2017-06-08; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Caries Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors will not be blind to intervention/control assessment methods. However it will not be allowed amongst the examiners to exchange any information throughout the entire study period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICDAS (Active Comparator): International Caries Detection and Assessment System : Caries assessment system which is used to assess Any carious lesions then they are rated in codes from 0,1,2,3,4,5,6
  Interventions: Diagnostic Test: International Caries Classification and Management System
- ICCMS (Experimental): International Caries Classification and Management System Any carious lesions detected are rated in score as the follow:Code 0 = ICDAS 0 Code A = ICDAS 1,2 Code B = ICDAS 3,4 Code C= ICDAS 4,6
  Interventions: Diagnostic Test: International Caries Classification and Management System

INTERVENTIONS:
Diagnostic Test: International Caries Classification and Management System — Caries assessment and management system
  Other Names: ICCMS

SUMMARY:
1. A total of 40 volunteer patients will be assigned in this study.
2. All patients will be randomly selected with variable caries risks .
3. For each patient The Examiner will use Two screening methods used in caries detection , where D1 represents ICDAS index and D2 represents ICCMS index which are used by each examiner for each patient.
4. Each examiner will record the dental findings using the visual- tactile assessment method .The visual-tactile assessment method includes the use of mirror, probe under good illumination condition
5. After full caries assessment in the 1st visit , All patients will receive full treatment and oral hygiene control .
6. After 6-months follow up re-assessment of same patients will be done by same Examiners .
7. The data of each examiner will be collected, and then the repeat-ability and the reproducibility of each method as well as the inter- and intra-operator agreement will be evaluated using the kappa statistics

   * Number of visits & follow up period: There will be 2 visits and 6-months follow up between 2 visits.
   * Direct benefit of the research to the human volunteer:To get the most appropriate treatment plan .
   * Scientific Value and social benefits:obtain better information quality and support Dentist Discussion making.
   * Expected risk to human subjects:: the ordinary side effects associated with any restorative treatment and no of the study variable has side effect on the patient and in case of any side effect due to the restorative treatment , the participant will directly contact the operator.

DETAILED DESCRIPTION:
1. Study setting ----------------------------- The study will be conducted in Conservative Dentistry Department, Faculty of Dentistry, Cairo University, The operator in charge will be: Amr Sobhy Abd Elmounem The researcher will bear ultimate responsibility for all activities associated with the conduct of a research project including recruitment of patients, explaining and performing the procedures to them
2. Variables of the study

   ------------------------------------

   A total of 40 volunteer patients will be assigned in this study. For each patient Two screening methods will be used in caries detection , where D1 represents ICDAS index and D2 represents ICCMS index which are used by each examiner for each patient
3. Intervention/control assessment:

   ------------------------------------------- Each examiner will record the dental findings using the visual- tactile assessment method .The visual-tactile assessment method includes the use of mirror, probe under good illumination condition.

   a. Control assessment: ICDAS

   Any carious lesions detected are rated in score as the follow:

   Code 0 Code 1 Code 2 Code 3 Code 4 Code 5 Code 6 .b. Intervention assessment: (International Caries Classification and Management System):

   Any carious lesions detected are rated in score as the follow:

   Code 0 = ICDAS 0 Code A = ICDAS 1,2 Code B = ICDAS 3,4 Code C= ICDAS 4,6
4. Outcome assessment:

   ---------------------------------- Each examiner will record the dental findings using both the intervention and control assessment method. Each method will be repeated twice at the first visit and the other after 6 months after oral hygiene control to calculate the repeat ability and reproducibility after and before treatment. The data of each examiner will be collected, and then the repeatability and the reproducibility of each method as well as the inter- and intra-operator agreement will be evaluated using the kappa statistics.
5. Participant timeline:

   ------------------------------ All procedures will be carried out in two visits
6. Sample size calculation:

   ---------------------------------- A sample size of 40 subjects achieves 80% power to detect an estimated Kappa value of 0.40; this power calculation is based on significance level 5%. The sample size was calculated by PASS 2008
7. Recruitment & Recruitment Strategy:

   -------------------------------------------------- Screening of patients that come to the conservative dentistry department seeking dental care will continue until the target population is achieved. The patients 'Oral condition will be subjected to visual examination and diagnosis using dental charts. Once the patients that are potentially eligible for this study are identified, they will be contacted by the research investigator who will explain the study and ascertains the patient's interest. If interested, more detailed evaluations and preparations are made.
8. Randomization and assignment of interventions:

   --------------------------------------------------------------- No randomization will be done as all patients will be examined by all examiners

   Blinding:

   The assessors will not be blind to intervention/control assessment methods. However it will not be allowed among the examiners to exchange any information throughout the entire study period.
9. Data collection methods:

   ---------------------------------- Caries will be assessed by both methods. Patients with other dental work, not included in the study design, will be treated prior to recruitment. Examiners will record the dental findings of the diagnosed fillings by both intervention/control assessment methods on a dental chart.
10. Data management:

    --------------------------- The data will be entered and stored on a personal computer. Double data entry will be saved on an external hard disc to prevent loss of data
11. Statistical methods:

    -------------------------------- Data will be analyzed using advanced statistics IBM SPSS . Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages. Correlation analysis will be used. Agreement between both methods will be analyzed with the use of kappa statistics
12. Monitoring:

    --------------------- A. Data monitoring: The main supervisor will monitor this study. His role is to monitor any risk of bias could be done from participants

    B. Harms:

    The main researcher should inform participants about the possible harms, if present. Participants are allowed to contact the main researcher at moment through telephone

    C. Auditing:

    In the present trial, auditing will be done by the main and co-supervisors to assure quality of the research frequency procedures

13-Ethics and Dissemination:

1. Research ethics approval:

   Application forms for carrying out the clinical trial, checklist and informed consent of Research Ethics Committee (REC) Faculty of Oral and Dental Medicine, Cairo University will be retrieved and filled, then will be delivered for (REC) committee for approval. This is done to prevent any ethical problems during the study or any harm for any of the participants.
2. Protocol amendments:

   If a new protocol will be used a protocol amendment will be submitted; containing a new copy of the new protocol and brief explanation about the differences between it and the previous protocols. If there is a change in the existing protocol that affects safety of subjects, investigation scope or scientific quality of the trial, an amendment containing a brief explanation about the change will be submitted. If a new author will be added to accomplish the study, an amendment including the investigator's data and qualifications to conduct the investigation will be submitted to prevent ghost authorship.
3. Consent:

   The operator (Amr sobhy Abd elmounem) is responsible for admitting and signing the written consents during the enrollment day.
4. Confidentiality:

   Name, personal data and pictures of the participants will not appear on the protocol form and will be maintained secured for 10 years after the trial. This is done for protection of participants' privacy and civil rights.
5. Declaration of interests:

   There is no conflict of interest, no funding or material supplying from any parties.
6. Access to data:

   Access to final data will be allowed to the operator, the main and co-supervisors of the study who are not involved in assessment of the outcome.
7. Dissemination policy:

Full protocol will be published online in www.clinicaltrials.gov to avoid repetition and to keep the integrity of the research work. Thesis will be discussed in front of judgment committee. The study will be published to report the results of this clinical trial.

14. Dissemination policy:

------------------------------- Full protocol will be published online in www.clinicaltrials.gov to avoid repetition and to keep the integrity of the research work.Thesis will be discussed in front of Judgment committee. The study will be published to report the results of this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Articles published in English
* Articles published after 2002.
* ICDAS & ICCMS
* Reproducibility

Exclusion Criteria:

* In any other languages.
* Articles published before 2002.
* Any other clinical evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-03 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Validity of screening system | an average of 1 year
  The outcome( Validity) will be measured by measuring Reproducibility of each screening system using Kappa equation .

CONTACTS AND LOCATIONS:
Overall Officials: omima Safwat, PHD, Study Director — Professor of Conservative Dentistry, Cairo University; Amir Hafez, PHD, Study Chair — Lecturer of Conservative Dentistry, Cairo University
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes